CLINICAL TRIAL: NCT00003446
Title: Phase II Trial of Trimetrexate (Neutrexin), 5-Fluorouracil and Leucovorin in Metastatic Colorectal Cancer
Brief Title: Chemotherapy in Treating Patients With Recurrent or Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Oncologico Cooperativo del Sur (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: GOCS-12-CR-97; CDR0000066475 (Registry Identifier: PDQ (Physician Data Query)); NCI-V98-1457
Record Dates: First submitted 1999-11-01; First posted 2004-04-09 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2001-09

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Fluorouracil; Leucovorin; trimetrexate glucuronate

INTERVENTIONS:
Drug: fluorouracil
Drug: leucovorin calcium
Drug: trimetrexate glucuronate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of trimetrexate glucuronate, fluorouracil, and leucovorin in treating patients with recurrent or metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate tumor response and duration, one-year progression-free survival, and one-year overall survival in patients with recurrent or metastatic colorectal carcinoma when treated with trimetrexate glucuronate, fluorouracil, and leucovorin calcium.

OUTLINE: Patients receive trimetrexate glucuronate (TMTX) IV over 1 hour on day 1. Beginning 18 hours after the TMTX dosage, patients receive leucovorin calcium (CF) IV over 2 hours. Immediately after the completion of the CF infusion, patients receive an IV bolus injection of fluorouracil (5-FU). Beginning 4 hours after the 5-FU infusion, patients receive oral CF every 6 hours for 6 doses. Treatment repeats every 14 days in the absence of disease progression or unacceptable toxicity or as long as the disease remains inoperable. Patients are followed every 3 months for 1 year, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 18-45 patients will be accrued for this study within 15 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed colorectal carcinoma Inoperable advanced recurrent or metastatic disease Measurable disease outside previously irradiated area No CNS metastases

PATIENT CHARACTERISTICS: Age: 18 to 74 Performance status: WHO 0-1 Life expectancy: More than 12 weeks Hematopoietic: WBC greater than 4,000/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin less than 1.25 times upper limit of normal (ULN) SGOT less than 1.25 times ULN Albumin greater than 3.5 g/dL Renal: Creatinine clearance greater than 70 mL/min Cardiovascular: No history of congestive heart failure, myocardial infarction within the past 6 months, active ischemic heart disease, or uncontrolled hypertension Other: No weight loss more than 10% in the last 2 months No other prior malignancy except curatively treated carcinoma in situ of the cervix or non-melanoma skin cancer No history of alcohol abuse No uncontrolled medical or psychiatric disease Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent filgrastim (G-CSF) Chemotherapy: No prior chemotherapy for advanced disease Recovered from prior adjuvant therapy No other concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics No prior radiotherapy for advanced disease Surgery: See Disease Characteristics Other: No other concurrent therapy

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1997-12; Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan Eduardo Perez, MD, Study Chair — Grupo Oncologico Cooperativo del Sur
Locations (1):
- Grupo Oncologico Cooperativo del Sur, Bahía Blanca, Buenos Aires, Argentina